CLINICAL TRIAL: NCT02301949
Title: The Study of the Optimal Treatment Strategy for Patients With Gastrointestinal Bleeding Due to Gastrointestinal Vascular Malformation: a Randomized, Double Blind, Placebo Controlled Study
Brief Title: Retreatment and Its Efficiency of Thalidomide for Vascular Malformation Patients With Failure of First Course Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Zhizheng Ge (Other)
Responsible Party: Sponsor-Investigator, Zhizheng Ge, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjyyxhnj3015
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Gastrointestinal Bleeding of Unknown Origin; Gastrointestinal Vascular Malformation; Thalidomide Efficiency
Keywords: gastrointestinal bleeding; vascular malformation; thalidomide retreatment
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Vascular Malformations | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thalidomide Retreatment Group (Active Comparator)
  Interventions: Drug: Thalidomide
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Thalidomide — Patients are randomly assigned to receive a second course of four-month treatment of thalidomide (Pharmaceutical Co., Ltd. of ChangZhou, China). Medications are taken orally 25mg four times daily at 6 a.m., 12 noon, 6 p.m., and 10 p.m.
  Other Names: Softenon
  Arms: Thalidomide Retreatment Group
Other: Placebo — Patients are randomly assigned to receive placebo tablets (Pharmaceutical Co., Ltd. of ChangZhou, China) four times daily at 6 a.m., 12 noon, 6 p.m., and 10 p.m.
  Arms: Placebo Group

SUMMARY:
Background: Repeated episodes of bleeding from gastrointestinal vascular malformations refractory to endoscopic or surgical therapy often pose a major therapeutic challenge.

Methods: The investigators will perform a randomized, double blind, placebo controlled study of thalidomide as a retreatment therapy for recurrent gastrointestinal bleeding due to vascular malformation. Patients with failure of first course treatment of thalidomide will be randomly grouped, prescribed a second four-month course regimen of 25 mg of thalidomide or placebo orally four times daily. All patients will be monitored for at least one year. The primary end point is defined as the patients whose rebleeds decrease from baseline by ≥ 50% at 12 months and the cessation of bleeding. Rebleeding is defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment. Secondary outcomes include the participants dependent on blood transfusions and changes from baseline in transfused packed red cell units, bleeding episodes, and hemoglobin levels at 12 months. Statistical significance is defined at P < 0.05.

DETAILED DESCRIPTION:
Protocol Description:

This is an exploratory, randomized, double blind, placebo controlled study of thalidomide for retreatment patients with failure of first course thalidomide treatment for recurrent gastrointestinal bleeding from vascular malformations. Informed consent will be taken from all subjects and the Institute Ethics Committee approved the study protocol. All procedures are in accordance with the Declaration of Helsinki. The study is not supported by pharmaceutical funding.

Study design and Intervention:

From Dec. 2014 to Nov. 2015, patients with failure of first course thalidomide treatment and repeated at least four episodes of chronic gastrointestinal bleeding a year due to vascular malformations identified by oesophagogastroduodenoscopy, capsule endoscope or double-balloon endoscope will be enrolled (according our enrollment criteria).

The patients will be randomly assigned to receive a second four-month course of 25 mg of thalidomide or placebo at daily time 6 a.m.,12 noon,6 p.m. and 10 p.m., respectively.

Randomization is performed through the proc plan procedure of Statistical Analysis System (SAS), using the method of randomly permuted blocks of 4. Within each block, the number of patients allocated to each of the two treatments is equal. Each patient who met the inclusion criteria will be consecutively assigned a random number in chronological order, which allocate him or her to one of the treatment groups.

In the case of an adverse event, the study medication will be temporarily or permanently discontinued based on subject inclination and toxicity intolerance.

Concomitant therapies, such as blood transfusions and other symptomatic treatments like iron supplementation, will be performed in both groups as necessary during the four-month treatment and subsequent follow-up periods. Blood transfusion is indicated and recorded when the hemoglobin (Hb) level reaches < 7.0 g/dl. Red-cell transfusions are administered according to patient Hb level as follows: 2 units will be administered for 6.1 g/dl ≥ Hb ≤ 7.0 g/dl, 3 units for 5.1 g/dl ≥ Hb ≤ 6.0 g/dl, and 4 units for Hb < 5.0 g/dl. Iron is provided for patients with 7.0 g/dl ≥ Hb ≤ 11.0 g/dl. After the four-month treatment course, all patients discontinued study medications except for cases where symptomatic treatments are necessary as described above.

Assessment of response and adverse events:

The primary end point is defined as the patients whose rebleeds decrease from baseline by ≥ 50% at 12 months and the cessation of bleeding. Rebleeding is defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment. Secondary outcomes include the participants dependent on blood transfusions and changes from baseline in transfused packed red cell units, bleeding episodes, and hemoglobin levels at 12 months.

Adverse events include any unfavorable change in health, including abnormal laboratory findings, during the study or follow-up period.

Evaluation of Patients and Follow-up:

* Certified research nurses collected information on the demographics and medical and social histories of all patients enrolled in the study.
* After screening and baseline evaluations, the patients will be closely monitored in the hospital for at least one week. They are then followed twice monthly during the four-mouth course of treatment and once a month thereafter.
* Clinical follow-up is performed by qualified doctors. At all visits, the bleeding-related parameters (number and duration) will be collected, a physical examination will be performed and laboratory values obtained for FOBT, complete blood counts, serum chemistries, and hepatic and renal function. Neuropathy and other adverse events were also assessed.
* Patients are advised to refrain from any other non-prescribed medicines, especially rebleeding-related medications such as aspirin, nonsteroidal anti-inflammatory drug(NSAIDs), anti-platelet drugs, anticoagulants, and Chinese medications (with salicylates), gingko, or Echinacea.

Statistical Analysis:

To our knowledge, no similar such study concern on efficiency of thalidomide retreatment has previously been performed, and the investigators are thus unable to refer to published studies to determine our samples. According to our published study, response in the iron-control group and thalidomide group reached 3.7% and 71.4%. And in our preliminary study (unpublished), response of thalidomide retreatment reached 66.7%. For this study, the investigators estimate that the primary outcome (the proportion of subjects whose number of yearly bleeds has decreased by ≥ 50%) will occur in 3.7% of the placebo group and 66.7% of the thalidomide retreatment group patients. An equally divided sample of 9 subjects is deemed sufficient for detecting the primary end point, with a type I error (two-sided) of 5% and a power of 90%. Assuming a 10% volunteer attrition rate to follow-up, the investigators establish a target sample size of 10 per group (calculated with PASS 11). To ensure an adequate power of later stratified analysis, the sample size is approximately increased to be 15 in each group.

Analyses of the responses and adverse events are performed on all registered patients according to the intention-to-treat principle. Statistical analysis is performed by a blinded biostatistician with the SPSS 13.0 software package. The investigators simultaneously analyze the primary endpoint of the full analysis set (FAS) and per protocol set (PPS). Continuous variables are compared using a two-sample independent t-test or Wilcoxon rank-sum test. Categorical variables are compared using the chi-squared and Fisher's exact tests. The Breslow-Day test is used to test for the heterogeneity of treatment effects across strata. All reported P-values are two-sided. Data are reported as the mean ±Standard Deviation(SD) or median (range) for continuous variables and number (%) for categorical variables. Since adjustments to the control group are minimal, the investigators also report point estimates and 95% confidence intervals (CIs). For all outcomes, a P-value of < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-85 years; women are post-menopausal, post-tubal ligation, or on some form of birth control like long-term laying up contraceptive ring or using condom;
* Patients with failure of first course treatment of thalidomide, which means rebleeds decreased from baseline by< 50% at 12 months follow up ;
* History of at least six documented gastrointestinal bleeding episodes in the year prior first course thalidomide treatment, which are refractory or inaccessible to endoscopic therapy or surgical ectomy; so, patients should have at least four episodes of gastrointestinal bleeding a year prior our study;
* Confirmed diagnosis of vascular malformation by esophagogastroduodenoscopy (EGD), capsule endoscope (CE), double-balloon endoscope (DBE), or colonoscopy, but no obvious infectious, neoplastic, or other specific diagnosis;
* Angiodysplasia at endoscopy characterized by focal or diffused venous/capillary lesions presenting as bright red ectatic vessels or pulsatile red protrusions, with surrounding venous dilatation or patchy erythema with or without oozing;
* Endoscopic appearance of GAVE (also known as watermelon stomach), indicated by longitudinal antral folds converging on the pylorus, containing visible columns of tortuous red ecstatic vessels.

Exclusion Criteria:

* Patients are excluded if first course treatment of thalidomide is effective, which means rebleeds decreased from baseline by ≥ 50% at 12 months follow up;
* if they have cirrhotic or portal hypertension gastropathy; severe co-morbidities of cardiac, pulmonary, renal, liver, hematological, rheumatologic disorders, or uncontrollable diabetes mellitus or hypertension;
* if they have a history of severe bilateral peripheral neuropathy or seizure activity, thromboembolic disease, known thalidomide allergy;
* if they have a history of treatment with any dose of systemic or oral topical corticosteroids or aspirin, NSAIDs, anti-platelet drugs, anticoagulants, or Chinese medications (with salicylates), gingko, or Echinacea, or other putative immunomodulators or anti-angiogenic agents;
* Currently pregnant or lactating or currently undergoing systemic cancer chemotherapy or receiving radiation

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point is defined as the patients whose rebleeds decrease from baseline by ≥ 50% at 12 months | 12 months
  The primary end point is defined as the patients whose rebleeds decrease from baseline by ≥ 50% at 12 months. Reduction of rebleeds = [(total bleeding episode at 12 months - total bleeding episodes at a year before randomization)/total bleeding episodes at a year before randomization(baseline)]*100%. Rebleeding is defined based on a positive fecal occult blood test (FOBT) (monoclonal colloidal gold color technology) at any visit after treatment.

SECONDARY OUTCOMES:
Change From Baseline in Hemoglobin (Hb) Level at 12 Months | 12 months
  The change from baseline in average hemoglobin (Hb) level(tested every month) at 12 months.
Change From Baseline in Bleeding Episodes at 12 Months | 12 months
  The Change from baseline in bleeding episodes at 12 months
Participants Dependent on Blood Transfusions | 12 months
  Numbers of participants dependent on blood transfusions
Change From Baseline in Total Transfused Red Cell Requirements at 12 Months | 12 months
  Change of total transfused red cell requirements at 12 months after randomization from one year before baseline in transfusion dependent patients
Cessation of Bleeding | 12 months
  The cessation of bleeding is defined as repeated negative faecal occult blood test (FOBT) (monoclonal colloidal gold color technology) during our observation period. Rebleeding is defined based on a positive FOBT at any visit after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhizheng Ge, MD. Ph.D, Principal Investigator — Shanghai Ren Ji Hospital
Locations (1):
- Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Jacobson JM, Greenspan JS, Spritzler J, Ketter N, Fahey JL, Jackson JB, Fox L, Chernoff M, Wu AW, MacPhail LA, Vasquez GJ, Wohl DA. Thalidomide for the treatment of oral aphthous ulcers in patients with human immunodeficiency virus infection. National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group. N Engl J Med. 1997 May 22;336(21):1487-93. doi: 10.1056/NEJM199705223362103. PMID 9154767
- [Background] Bauditz J, Schachschal G, Wedel S, Lochs H. Thalidomide for treatment of severe intestinal bleeding. Gut. 2004 Apr;53(4):609-12. doi: 10.1136/gut.2003.029710. PMID 15016759
- [Background] Shurafa M, Kamboj G. Thalidomide for the treatment of bleeding angiodysplasias. Am J Gastroenterol. 2003 Jan;98(1):221-2. doi: 10.1111/j.1572-0241.2003.07201.x. No abstract available. PMID 12526972
- [Background] Ge ZZ, Chen HM, Gao YJ, Liu WZ, Xu CH, Tan HH, Chen HY, Wei W, Fang JY, Xiao SD. Efficacy of thalidomide for refractory gastrointestinal bleeding from vascular malformation. Gastroenterology. 2011 Nov;141(5):1629-37.e1-4. doi: 10.1053/j.gastro.2011.07.018. Epub 2011 Jul 22. PMID 21784047